CLINICAL TRIAL: NCT01937429
Title: GRAND BLEU Study: Does the Colonoscopy With Instillation of Blue Water (Indigo Carmin® Dilute) Enable an Improved Rate of Adenoma Detection for Colonoscopy With Insufflation of Air?
Brief Title: Effectiveness of Instillation of Blue Water (Indigo Carmin®) for Colonoscopy
Acronym: GRAND BLEU
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012.713
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Adenoma Detection to Prevent Colorectal Cancer
Keywords: Colonoscopy - Chromoendoscopy - Indigo Carmin® - Adenoma detection - Tepid water
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colonoscopy with blue indigo Carmin® (Experimental): Patients undergoing from a colonoscopy with instillation of tepid water (30°C) tinged with indigo Carmin® (0,08/1000) during the endoscope insertion from the anus to the caecum, and with insufflation of air only during withdrawal from the caecum to the anus.
  Interventions: Device: Colonoscopy with blue Indigo Carmin®
- Standard colonoscopy (Active Comparator): Standard colonoscopy with insufflation of air
  Interventions: Device: Standard colonoscopy with insufflation of air

INTERVENTIONS:
Device: Colonoscopy with blue Indigo Carmin®
  Arms: Colonoscopy with blue indigo Carmin®
Device: Standard colonoscopy with insufflation of air
  Arms: Standard colonoscopy

SUMMARY:
The colonoscopy is the reference examination for the diagnosis of neoplastic lesions in the colon and rectum. Mass screening assessment studies have shown that colonoscopic detection and removal of adenomas in patients selected through fecal occult blood test reduces colorectal cancer incidence and mortality. However, the literature has reported interval cancer cases or adenomas, probably "missed" by the colonoscopy. In theory, using coloured warm water could improve colon preparation by mobilizing the residual faeces, decreasing the colic spasm and increasing the visualization of the pit pattern. Preliminary American studies, led by Leung et al, have shown a very clear increase in the adenoma detection rate.

The investigators' study involves 1 000 patients, treated in the Rhône-Alpes / Auvergne region. The patients present an indication for colonoscopy following a positive fecal occult blood test or symptoms or personal and family histories of pre-cancerous colonic lesions. They will be randomized into two study groups:one of both groups of study: Group 1: patients undergoing a colonoscopy wtih instillation of tepid water tinged with blue (Indigo Carmin®) Group 2: patients undergoing a standard colonoscopy with insufflation of air. The main objective is to show that the colonoscopy with blue water (Indigo Carmin®) enable detection of more lesions than standard colonoscopy with insufflation of air. The two techniques will be also compared in terms of tolerance, of duration of colonoscopy and type of detected lesions.

In case of improved detection of colorectal lesions, the blue water instillation technique of could dramatically change gastroenterologists' practice by becoming the reference method. The expected clinical benefits are potential revealing of more neoplastic lesions and improvement in abdominal discomfort after colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older
* Scores 1 to 3 in ASA (American Society of Anesthesiologists) classification
* Patient having an indication for of colonoscopy to detect colorectal neoplastic lesions, which meet at least one of the following conditions:

  * Positive fecal occult blood Test
  * 1st degree family history of colorectal cancer or adenoma before 60 years of age
  * Personal history of colorectal adenomas or colorectal cancer
  * Unexplained digestive symptoms after 50 years of age or those not responding to symptomatic treatment: modification of bowel movements, abdominal pains
  * Isolated or repeated rectal bleeding after 50 years of age or occult bleeding
  * Acromegaly
  * Infectious endocarditis with digestive bacteria
* No coagulation anomalies or no taking of medicine affecting coagulation
* Signing of informed consent form before the performance of any procedure related to the study

Exclusion Criteria:

* Known inflammatory or infectious colorectal disease
* Hereditary Non Polyposis Colorectal Cancer disease (Lynch syndrome) or family history of adenomatous polyposis
* Histories of colorectal surgical resection
* Known hypersensitivity to indigo Carmin® or to one of the preparation components
* Pregnant or breastfeeding women, or those likely to become pregnant without effective contraception
* patient not affiliated with a social security care system or who do not benefit from such a system
* Patient over 18 years of age protected by the Law, under guardianship or curators
* Concomitant participation in an interventional biomedical research trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
The rate of colonoscopy with at least one adenoma detected (or adenoma detection rate) confirmed by a histological reporting. | Within the first 20 days after colonoscopy.

SECONDARY OUTCOMES:
Measure 1: The characteristics of the lesions detected by the two types of colonoscopy (diameter, macroscopic appearance, histological nature) | within the first 20 days after colonoscopy.
  We chose three classifications recognized by the medical field:
  1. The Paris endoscopic classification defines macroscopic appearance.
  2. The Kudo classification explains endoscopic appearance.
  3. The Vienna classification describes the histologic nature of the lesions.
Measure 2 Comparison of the time of the endoscope during the colonoscopy between the two methods | This data is available during the colonoscopy
Measure 3 The comparison of the tolerance of the two colonoscopy procedures by assessing patient reported side effects. | At patient's awakening the day of colonoscopy or one day after
  Tolerance is measured using a Visual Analog Scale.
  The questionnaire includes four questions :
  * Did you have any pains?
  * How would you describe your bloating?
  * How would you describe your sensations of abdominal discomfort?
  * How would you describe your overall tolerance of the examination?
  In addition to this Visual Analog Scale, we administer a short multiple choice questionnaire:
  * Would you be ready to redo the colonoscopy in the same conditions? (yes or no)
  * For patients who have already had colonoscopies with insufflation of air in the past, which examination (tepid water or air) would you prefer during the next exam?

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PONCHON, MD, Principal Investigator — Hôpital E. Herriot -Service d'hépato-gastroentérologie
Locations (1):
- Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Derived] Lesne A, Rouquette O, Touzet S, Petit-Laurent F, Tourlonias G, Pasquion A, Rivory J, Aguero Garcete G, Scanzi J, Chalumeau S, Chambon-Augoyard C, Moussata D, Leger-Nguyen F, Degeorges S, Chauvenet M, Fontanges T, Baubet S, Brulet P, Billioud C, Thimonier E, Stroeymeyt-Martin K, Hamel B, Graillot E, Cruiziat C, Scalone O, O'Brien M, Pere-Verge D, Souquet JC, Phelip JM, Poincloux L, Poupon-Bourdy S, Denis A, Magaud L, Ponchon T, Pioche M. Adenoma detection with blue-water infusion colonoscopy: a randomized trial. Endoscopy. 2017 Aug;49(8):765-775. doi: 10.1055/s-0043-105073. Epub 2017 Apr 11. PMID 28399611